CLINICAL TRIAL: NCT01561911
Title: A Phase I Clinical Research Study Evaluating the Safety, Tolerability and Biological Effects of the Chimeric Anti-CD40 Monoclonal Antibody Chi Lob 7/4 Given Intravenously, Weekly for Four Weeks in the Treatment of Patients With Advanced Malignancies Refractory to Conventional Anti-cancer Treatment.
Brief Title: A Phase I Study of the Chimeric Anti-CD40 Monoclonal Antibody ChiLob 7/4 to Treat Advanced Malignancies Refractory to Conventional Anti-cancer Treatment
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Cancer Research UK (Other)
Responsible Party: Sponsor
Masking: None
Other Study IDs: PH1/103
Record Dates: First submitted 2012-03-21; First posted 2012-03-23 (Estimated); Last update posted 2014-12-02 (Estimated); Status verified 2014-12

CONDITIONS: Cancer; Neoplasms; Lymphoma; Non-Hodgkin; B-Cell
Keywords: Clinical Trial; Phase I; Antibodies; Monoclonal
MeSH Terms: conditions — Neoplasms; Lymphoma

INTERVENTIONS:
Drug: Chi Lob 7/4 (A chimeric monoclonal antibody) — 3 patients will receive treatment at each dose level. Escalation from one treatment dose level to another will only be permitted once at least 3 patients have completed treatment without any DLTs. Starting weekly dose of Chi Lob 7/4 will be 0.5mg (giving a total dose per patient of 2mg divided over 4 weeks). Subsequent individual, weekly dose levels of 1.6mg, 5mg, 16mg, 50mg and 160mg (resulting in total patient doses of 6.4mg, 20mg, 64mg 200mg and 640mg respectively). Further dose escalation can continue to 240mg and 320mg dose per week (resulting in 960mg and 1280mg. Patients may be treated at a lower or intermediate dose level to define the MTD/BAD.

SUMMARY:
The Purpose of this study is to evaluate the safety and tolerability, and the biological effects of the chimeric anti-CD40 monoclonal antibody Chi Lob 7/4, given intravenously, weekly for 4 weeks in the treatment of patients with advanced malignancies refractory to conventional anti-cancer treatment.

DETAILED DESCRIPTION:
The primary objective of the study is to establish the safety and maximum tolerated dose of Chi Lob 7/4. In line with other established antineoplastic, chimeric monoclonal antibody therapies such as Rituximab, Chi Lob 7/4 will be given by slow intravenous infusion once every week for a total of four weeks. This treatment regimen will facilitate early, rapid and dose dense administration of antibody to a patient group with advanced malignancy refractory to conventional treatment. The starting dose for each infusion of Chi Lob 7/4 will be 0.5mg (giving a total dose per patient of 2mg divided over 4 weeks). Escalation from one treatment dose level to another will only be permitted when at least 3 patients have completed treatment without dose limiting toxicity.

ELIGIBILITY:
Inclusion Criteria:

* Histologically proven CD40 expressing solid tumours or diffuse large B-cell non-Hodgkin"s lymphoma refractory to conventional treatment, or for which no conventional therapy exists.
* Written informed consent and the ability of the patient to co-operate with treatment and follow up must be ensured and documented.
* Age greater than 18 years.
* Life expectancy of at least 12 weeks.
* World Health Organisation (WHO) performance status of 0-1 (Appendix 1).
* Haematological and biochemical indices (These measurements must be performed within one week prior to the patient going on study.)

  * Haemoglobin (Hb) ≥ 9.0 g/dl
  * Neutrophils ≥ 1 x 10^9/L
  * Total Lymphocyte count ≥ 0.5 x 10^9/L
  * Platelets (Plts) ≥ 75 x 10^9/L
  * The following baseline liver function tests :

    * Serum bilirubin ≤ 1.5 x upper limit of normal (ULN)
    * Alanine amino-transferase (ALT) and/or aspartate amino-transferase (AST) ≤ 3 x ULN unless due to tumour in which case up to 5 x ULN is permissible
  * The following baseline renal function test:

    * calculated creatinine clearance ≥ 40 mL/min (uncorrected value) or isotope clearance measurement ≥ 40mL/min
* Female patients of child-bearing potential are eligible, provided they have a negative serum or urine pregnancy test prior to enrolment and agree to use appropriate medically approved contraception for four weeks prior to entering the trial, during the trial and for six months afterwards.
* Male patients must agree to use appropriate medically approved contraception during the trial and for six months afterwards.

Exclusion Criteria:

* CD40 negative tumours by immunohistochemistry.
* Radiotherapy (except for palliative reasons), endocrine therapy, immunotherapy or chemotherapy during the previous four weeks (six weeks for nitrosoureas and mitomycin-C) prior to treatment.
* All toxic manifestations of previous treatment must have resolved. Exceptions to this are alopecia or certain Grade 1 toxicities which in the opinion of the Investigator and Cancer Research UK should not exclude the patient.
* Pregnant and lactating women are excluded.
* Major thoracic and/or abdominal surgery in the preceding four weeks from which the patient has not yet recovered.
* Patients with primary brain tumours or clinically apparent brain metastases.
* Patients who are high medical risks because of non-malignant systemic disease including active uncontrolled infection.
* Patients with any other condition which in the Investigator"s opinion would not make the patient a good candidate for the clinical trial.
* Patients known to be serologically positive for Hepatitis B, Hepatitis C or Human Immunodeficiency Virus (HIV).
* Long term immunosuppression or steroids (for more than one month)
* History of significant and serious allergy.
* Concurrent congestive heart failure or prior history of class III/ IV cardiac disease (New York Heart Association [NYHA] - refer to Appendix 4)
* Patients with low grade or transformed non-Hodgkin"s lymphoma.
* Prior treatment with murine monoclonal antibodies. (Prior treatment with chimeric or fully human antibodies will not exclude a patient).
* A history of clinically significant autoimmune disease.
* Current malignancies at other sites, with the exception of adequately treated cone-biopsied in situ carcinoma of the cervix uteri and basal or squamous cell carcinoma of the skin. Cancer survivors, who have undergone potentially curative therapy for a prior malignancy, have no evidence of that disease for five years and are deemed at low risk for recurrence, are eligible for the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 29 (Actual)
Dates: Start 2007-07; Primary Completion 2014-10 (Actual); Study Completion 2014-10 (Actual)

PRIMARY OUTCOMES:
1. To establish the Maximum tolerated dose (MTD)of ChiLob 7/4 ;
  Defined as the dose below the dose at which no more 30% (2 of up to 6 patients in the cohort) , experienced a DLT (Dose Limiting Toxicity) due to ChiLob 7/4 occurring during the treatment period and up to 4 week's post treatment.
2. To determine the Biologically Active Dose of Chi Lob 7/4, which is defined as the dose level at which peripheral blood B-cells are reduced by the end of therapy to 10% or less of the starting number.
3. To determine the toxicity profile of Chi Lob 7/4 (CTCAE version 3.0) and to identify the dose limiting toxicity
4. To propose a safe dose for Phase II evaluation

SECONDARY OUTCOMES:
1. To examine the Biological effects of ChiLob 7/4 Treatment
2. To examine the Pharmacokinetics of ChiLob 7/4 treatment: (Measurement of Serum Chi Lob 7/4)
3. To examine the Possible Anti-Tumour activity of Chi Lob 7/4 (RECIST 1.0 criteria)

CONTACTS AND LOCATIONS:
Overall Officials: Peter W Johnson, Professor, Principal Investigator — Cancer Research UK Medical Oncology Unit, Southampton General Hospital,
Locations (2):
- United Kingdom (2):
  - Cancer Research UK Institute for Cancer Studies, University of Birmingham, Edgbaston, Birmingham
  - Cancer Research UK Medical Oncology Unit, Southampton General Hospital, Tremona Road,, Southampton

REFERENCES:
- [Derived] Johnson P, Challis R, Chowdhury F, Gao Y, Harvey M, Geldart T, Kerr P, Chan C, Smith A, Steven N, Edwards C, Ashton-Key M, Hodges E, Tutt A, Ottensmeier C, Glennie M, Williams A. Clinical and biological effects of an agonist anti-CD40 antibody: a Cancer Research UK phase I study. Clin Cancer Res. 2015 Mar 15;21(6):1321-8. doi: 10.1158/1078-0432.CCR-14-2355. Epub 2015 Jan 14. PMID 25589626
- See also: Click here for more information about the study: — http://cancerhelp.cancerresearchuk.org/trials/a-trial-looking-at-the-monoclonal-antibody-chi-lob-74-for-advanced-cancer